CLINICAL TRIAL: NCT01613859
Title: Measurement of Cardiac Output and Intravascular Volume Status in Critically Ill Children Using an Ultrasound Dilution Method (COstatus)
Brief Title: Measurement of Cardiac Output and Intravascular Volume Status in Children Using COstatus (SH)
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-COstatus-12A-H; R44HL061994 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2012-06-07 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Intensive Care

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Assessment and monitoring of cardiac function in the pediatric intensive care unit (PICU) is an integral part of hemodynamic monitoring of critically ill patients whether it is done directly or indirectly. Measurement of cardiac output (CO) can specifically guide therapies to support the cardiovascular system in critically ill children with multi organ dysfunction. Because of the side effects involved in measuring cardiac output directly, intensive monitoring of patients is currently limited to an integrated assessment of tissue perfusion, oxygen delivery and cellular health both at regional and global levels. Currently available methods of measuring CO have their limitations and complications, and are not used routinely for bedside monitoring. Therefore, the investigators propose to use a newly developed method, termed COstatus for the monitoring of CO in patients admitted to PICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients under 21 years
2. Presence of compensated or decompensated shock irrespective of etiology
3. Presence of an existing peripheral arterial and central venous catheters

Exclusion Criteria:

1. Patients allergic to heparin

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Patients (under 21 years of age) in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Comparing CO and other clinical markers in Pediatric ICU | During patients stay in ICU with insitu catheter, expected average 3-4 days
  The objective of this study is to see if the CO measurements obtained with COstatus show a linear correlation with all other indirect and invasive methods currently used to measure CO (within acceptable range) and with the CO measured by thermodilution in the cardiac catheterization lab.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Udassi, MD, Principal Investigator — Shands Children's Hospital, University of Florida
Locations (1):
- Shands Children's Hospital, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416